CLINICAL TRIAL: NCT03793309
Title: A Randomized Controlled Trial on the Effect of 400 vs. 800 IU of Vitamin D on T Regulatory Cells in Preterm Infants
Brief Title: Different Doses of Vitamin D and T Regulatory Cells in Preterm Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lamiaa Mohsen, professor of Pediatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12012016
Record Dates: First submitted 2018-12-24; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Prematurity; Immune Defect
MeSH Terms: conditions — Premature Birth | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental): Subjects in this group receive 400 IU vitamin D daily for 4 weeks.
  Interventions: Drug: Vitamin D
- High dose (Experimental): Subjects in this group receive 800 IU vitamin D daily for 4 weeks.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Oral vitamin D
  Other Names: Oral vitamin D

SUMMARY:
This study evaluate the effect of two different doses of vitamin D on T-regulatory cells in preterm infants. Half of the subjects receives 400 IU vitamin D and the other half receives 800 IU vitamin D.

DETAILED DESCRIPTION:
Vitamin D, in addition to its bone mineralization effect, is an immune- modulatory agent. Fetal and premature cellular immunity are generally delayed. Whether vitamin D can enhance cellular immunity by increasing T regulatory cells is unknown. The effect of two different doses of vitamin D; 400 IU and 800 IU will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age 28-33 weeks

Exclusion Criteria:

* Necrotizing enterocolitis
* Bowel perforation
* Chromosomal anomalies
* Inborn errors of metabolism
* Major congenital anomalies

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Percent Change in The Number of T Regulatory Cells | At 1 week (compared to baseline)
  Flow cytometry assessment of CD4+ , CD25+ with expression of FOXP3 will be used to identify T Regulatory cells
Percent Change in The Number of T Regulatory Cells | At 4 weeks (compared to baseline)
  Flow cytometry assessment of CD4+ , CD25+ with expression of FOXP3 will be used to identify T Regulatory cells

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Mohsen, MD, Principal Investigator — Cairo University Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bozkurt O, Uras N, Sari FN, Atay FY, Sahin S, Alkan AD, Canpolat FE, Oguz SS. Multi-dose vitamin d supplementation in stable very preterm infants: Prospective randomized trial response to three different vitamin D supplementation doses. Early Hum Dev. 2017 Sep;112:54-59. doi: 10.1016/j.earlhumdev.2017.07.016. Epub 2017 Aug 2. PMID 28779655
- [Result] Zittermann A, Dembinski J, Stehle P. Low vitamin D status is associated with low cord blood levels of the immunosuppressive cytokine interleukin-10. Pediatr Allergy Immunol. 2004 Jun;15(3):242-6. doi: 10.1111/j.1399-3038.2004.00140.x. PMID 15209957
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Aly H, Mohsen L, Bhattacharjee I, Malash A, Atyia A, Elanwary S, El Hawary R. Vitamin D Supplementation and T Cell Regulation in Preterm Infants: A Randomized Controlled Trial. J Pediatr Gastroenterol Nutr. 2019 Nov;69(5):607-610. doi: 10.1097/MPG.0000000000002448. PMID 31335838